CLINICAL TRIAL: NCT04590742
Title: Randomized Trial Investigating Melatonin Supplementation vs Placebo on Sleep Disturbance Following Total Joint Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JJP17D.511
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Sleep Disturbance; Total Joint Arthroplasty
MeSH Terms: conditions — Parasomnias | interventions — Melatonin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Placebo Comparator): Placebo Tablet
  Interventions: Drug: Placebo
- Group 2 (Active Comparator): Melatonin (6mg)
  Interventions: Drug: melatonin 6mg

INTERVENTIONS:
Drug: melatonin 6mg — 6 weeks of melatonin (6mg) given to patient
  Arms: Group 2
Drug: Placebo — Patient given 6 weeks of placebo tablet
  Arms: Group 1

SUMMARY:
The purpose of this study is to determine whether melatonin when used as a supplement after surgery improves sleep following total joint arthroplasty

ELIGIBILITY:
Inclusion Criteria:

1. Patients who undergo unilateral primary total joint arthroplasty
2. Patient willing and able to complete postoperative surveys

Exclusion Criteria:

1. Patients who undergo revision total joint arthroplasty
2. Patients who undergo bilateral total joint arthroplasty
3. Patients currently taking melatonin supplementation
4. Patient has history of substance abuse (drug or alcohol)
5. Patient is a workman's comp patient or patient has current litigation pending
6. Patient has an allergy to melatonin
7. Patient has a history of delirium/psychiatric/depression/on antidepressants
8. Patient has a history of insomnia/ on sleep aid medication
9. Anyone on warfarin
10. Sleep apnea
11. Patient discharged to SNF or rehab
12. Patients who have inflammatory conditions
13. Shift work or night work

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Patient Sleep Quality | 6 weeks
  Patients quality of sleep will be analyzed by having them answer a sleep quality index (PSQI) questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States